CLINICAL TRIAL: NCT00920244
Title: Dynamics and State Transitions During Resuscitation in In-hospital Cardiac Arrest
Brief Title: In-hospital Cardiac Arrest - Dynamics and State Transitions
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian Air Ambulance Foundation (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 4.2008.2402 (REK); 08/11457 (Other: SHDir); 20708/2/IB (Other: NSD)
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Heart Arrest; Death, Sudden, Cardiac
Keywords: Resuscitation; Cardiac arrest; State-transitions; Markov
MeSH Terms: conditions — Heart Arrest; Death, Sudden, Cardiac | interventions — Cardiopulmonary Resuscitation; Epinephrine; Atropine; Amiodarone; Defibrillators

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Cardiopulmonary resuscitation (CPR) — CPR is performed according to international and national guidelines on all patients.
  Other Names: CPR
Drug: Epinephrine — According to guidelines epinephrine 1 mg i.v. is administered every 3 minutes during cardiopulmonary resuscitation.
  Other Names: Adrenaline
Drug: Atropine — According to CPR guidelines atropine 3 mg i.v. is administered if asystole og PEA with frequency < 60 beat/min.
Drug: Amiodarone — According to guidelines amiodarone 300 mg i.v. is administered if recurrent ventricular fibrillation/tachycardia (VF/VT) during CPR.
  Other Names: Cordarone
Device: External defibrillator — According to CPR guidelines patients with shockable rhythms may receive DC shocks. The defibrillator also stores physiological information regarding cardiac rhythm, pulse-oximetry, and end-tidal carbon dioxide (CO2) from endotracheal tube.
  Other Names: Defibrillator

SUMMARY:
The purpose of this study is to analyse transitions in cardiac rhythm and hemodynamic variables during resuscitation of patients with in-hospital cardiac arrest.

DETAILED DESCRIPTION:
In-hospital cardiac arrest carries a grave prognosis, with survival to discharge in the range of 15-20%. Key factors determining outcome include the presenting cardiac rhythm, aetiology, and early initiation of resuscitation. Some cardiac rhythms benefit from defibrillation (shockable rhythms). During resuscitation patients may switch between shockable and non-shockable rhythms, and may show signs of spontaneous circulation temporarily. Depending on rhythm and according to guidelines, patients receive direct current (DC) shocks (defibrillator) and/or i.v. adrenaline, atropine and amiodarone, which may affect state-transitions. We wish to make statistical analysis (time-series analysis, Markov modelling) of these state-transitions and variations in hemodynamic variables during resuscitation, related to CPR interventions and the cause of arrest. The cause of arrest will be determined based on chart records, interview with staff and autopsy if appropriate. One hypothesis is that differences in the patterns of state-transitions may reflect underlying aetiology, which may guide in future decision-making during resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with in-hospital cardiac arrest who are resuscitated

Exclusion Criteria:

* Younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with in-hospital cardiac arrest at St.Olavs Hospital (Trondheim, Norway) during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2009-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Survival to discharge | 1 year

SECONDARY OUTCOMES:
Short-term survival | minutes-days

CONTACTS AND LOCATIONS:
Overall Officials: Eirik Skogvoll, MD, PhD, Study Chair — St. Olavs Hospital; Trond Nordseth, MD, Principal Investigator — St. Olavs Hospital
Locations (1):
- St.Olavs Hospital, Department of Anesthesia, Trondheim, Norway

REFERENCES:
- [Result] Skjeflo GW, Nordseth T, Loennechen JP, Bergum D, Skogvoll E. ECG changes during resuscitation of patients with initial pulseless electrical activity are associated with return of spontaneous circulation. Resuscitation. 2018 Jun;127:31-36. doi: 10.1016/j.resuscitation.2018.03.039. Epub 2018 Apr 3. PMID 29621571
- [Derived] Nordseth T, Bergum D, Edelson DP, Olasveengen TM, Eftestol T, Wiseth R, Abella BS, Skogvoll E. Clinical state transitions during advanced life support (ALS) in in-hospital cardiac arrest. Resuscitation. 2013 Sep;84(9):1238-44. doi: 10.1016/j.resuscitation.2013.04.010. Epub 2013 Apr 19. PMID 23603153